CLINICAL TRIAL: NCT05637502
Title: Graded Motor Imagery in Women Diagnosed With Genito-Pelvic Pain Penetration Disorder. A Randomized Controlled Trial
Brief Title: Graded Motor Imagery in Women Diagnosed With Genito-Pelvic Pain Penetration Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Borja Pérez-Domínguez, Assistant Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UV-INV_ETICA-2678233
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Genito-Pelvic Pain/Penetration Disorder
Keywords: Genito-Pelvic Pain/Penetration Disorder; Pelvic pain; Dyspareunia; Graded Motor Imagery; Physical Therapy
MeSH Terms: conditions — Pelvic Pain; Dyspareunia

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graded Motor Imagery (Experimental): Participants receiving a tailored Graded Motor Imagery program for pelvic pain.
  Interventions: Other: Graded Motor Imagery
- Control (No Intervention): Participants initially receiving no intervention at all.

INTERVENTIONS:
Other: Graded Motor Imagery — Graded Motor Imagery programme consisting on three stages that will be gradually implemented. (i) Implicit Motor Imagery, that will be implemented through a developed app that resembles the Recognize app but adapted for Pelvic Floor disorders, (ii) Explicit Motor Imagery, applied through several sessions of motor imagery assisted through audio recordings and (iii) Graded Exposure, also guided through audio recordings and several practical tasks to perform.
  Arms: Graded Motor Imagery

SUMMARY:
The goal of this clinical trial is to assess the effects of a Graded Motor Imagery (GMI) programme in women diagnosed with Genito-Pelvic Pain Penetration (GPPD) Disorder.

The main questions it aims to answer are:

Does a GMI programme reduce pain intensity levels in women diagnosed with GPPPD? Does a GMI programme have an effect on sexual function in women diagnosed with GPPPD?

Participants will undergo a GMI programme and will be tested prior to and after the intervention to assess if the programme has a significant effect with regards to pain intensity and other pain-related outcome

DETAILED DESCRIPTION:
Graded Motor Imagery has been extensively used in several populations suffering pain-related disorders. It triggers cortical stimulation gradually in order to have an effect on the alterations that might have occured due to pain

Women suffering from Genito-Pelvic Pain Penetration Disorder deal with persistent pelvic pain that is no longer responding to a noxious stimulus, therefore this clinical presentation could have several cortical alterations implicated.

The main goal of this study is to assess if a Graded Motor Imagery programme is able to reduce pain intensity and improve sexual function in women diagnosed with Genito-Pelvic Pain Penetration Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with persistent pelvic pain
* Pain suffered for a period of a minimum of 3 months
* Adult (>18 years) women

Exclusion Criteria:

* Medical condition that logically explains the presence of pain
* Pain suffered for a period of less than 3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-22 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 6 weeks
  Pain intensity assessed through a Visual Analogue Scale, with a mininum value of 0 and a maximum value of 10, higher scores mean a worse outcome
Sexual function | 6 weeks
  Sexual function assessed through a short version of the Female Sexual Function Index (FSFI). Minimum score is 6, maximum score is 30. Higher scores mean better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No